CLINICAL TRIAL: NCT06818864
Title: Deep Brain Stimulation (DBS) for the Treatment of Cognitive Deficits After Traumatic Brain Injury (TBI): Pilot Trial
Brief Title: DBS for Cognitive Deficits After Traumatic Brain Injury
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Neurosurgeon, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5762
Record Dates: First submitted 2024-11-20; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: TBI Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: This is a phase I, non-blinded, non-randomized, open-label, pilot trial for safety and efficacy of deep brain stimulation for TBI. Patients who meet inclusion and exclusion criteria will be identified and recruited from the practices of psychiatrists and neurologists who specialize in treating patients with TBI who develop cognitive deficits. The study will proceed according to the schedule laid out below. Both patients and treating team will be aware of treatment parameters at all times. Up to ten (10) subjects will be enrolled. Study duration for each patient will be of one (1) year. Previous phase I trials of DBS in psychiatric populations have utilized 5-6 subjects per surgical target. Such a number has been sufficient to demonstrate initial safety, feasibility and provide preliminary data on clinical effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Patients will arrive on the morning of surgery to the medical imaging department of the Sunnybrook Hospital. They will have a stereotactic frame attached directly to their skull, after infiltration with local anesthesia. The frame allows precise coordinates to be acquired so that deep brain structures can be targeted with implanted electrodes. The patient will then undergo a CT scan with the frame in place, followed by transport directly to the operating room. The anesthesia team will insert an intravenous line and may use gentle sedation to relax the patient prior to and during the operation, as they will remain awake during the first stage of the operation. In the operating room the patient's head, via the frame, will be attached to the operating room table, and their scalp infiltrated with additional local anesthetic. A skin incision will be made and two burr holeswith approximately 1.4cm in diameter drilled through the skull. A small electrode will identify the optimal spot for el
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Patients will arrive on the morning of surgery to the medical imaging department of the Sunnybrook Hospital. They will have a stereotactic frame attached directly to their skull, after infiltration with local anesthesia. The frame allows precise coordinates to be acquired so that deep brain structures can be targeted with implanted electrodes. The patient will then undergo a CT scan with the frame in place, followed by transport directly to the operating room. The anesthesia team will insert an intravenous line and may use gentle sedation to relax the patient prior to and during the operation, as they will remain awake during the first stage of the operation. In the operating room the patient's head, via the frame, will be attached to the operating room table, and their scalp infiltrated with additional local anesthetic. A skin incision will be made and two burr holeswith approximately 1.4cm in diameter drilled through the skull. A small electrode will identify the optimal spot for ele

SUMMARY:
Patients with memory and cognitive deficits following TBI that do not respond to conventional treatments experience a decrease in quality of life. Despite advances in neuroimaging, genetics, pharmacology and psychosocial interventions in the last half century, little progress has been made in altering the natural history of the condition or its outcome.

This study would explore whether a surgical therapy is safe and potentially effective in patients who develop refractory memory and cognitive deficits following TBI. Preclinical studies suggest that DBS may improve memory deficits in TBI models. Moreover, DBS delivered to the fornix has shown promising clinical results in patients with Alzheimer's disease. The main mechanism for the improvements induced by DBS in memory tests is the development of multiple forms of plasticity.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a significant public health issue with an incidence of 55-70 million individuals worldwide. In Canada, TBI leads to 23,000 hospitalizations per year with 8% of individuals succumbing to their injuries. In addition to neurologic deficits, TBI may lead to a spectrum of long-term impairments, including cognitive difficulties (e.g., attention, memory), neurologic symptoms (e.g., headaches, dizziness) and neuropsychiatric sequalae (e.g. anxiety, post-traumatic stress disorder). TBI has also been associated with neurodegenerative disorders, such as chronic traumatic encephalopathy and the development of Alzheimer's-type pathology.

Cognitive rehabilitation programs are important tools for clinical recovery of TBI patients, improving functional outcomes and the quality of life. Some of these strategies are based on the development of compensatory strategies and neuroplasticity. Due to the short liver nature of some of the associated improvements and neuroplastic phenomena, stimulating specific neuronal circuits has been proposed.

To date, class I evidence suggests that cognitive improvement following rehabilitation is more effective than sham treatment. In general, however, cognitive rehabilitation therapy is effective in 80-90% of patients. This means that 10-20% of patients remain severely disabled despite treatment.

Deep Brain Stimulation is a neurosurgical tool that has been widely used for over twenty years. Most of the experience with DBS comes from the movement disorder literature where significant success has been had with the management of disabling Parkinson's Disease (PD) and dystonia. Owing to similar underlying circuitry, and the frequent co-occurrence of psychiatric and neurologic conditions, DBS has been suggested for the management of treatment resistant neuropsychiatric conditions, with some promising results.

To date, clinical studies using DBS following TBI are largely comprised of case reports and small case series. The most common application of invasive neurostimulation has been for the treatment of post-TBI dystonic symptoms and tremor. In addition to motor improvement, Miller et al reported a series of 4 patients who presented an improvement in visuospatial memory following fornix burst stimulation. Zhou et al reported that DBS delivered to the anterior limb of internal capsule and the region of the nucleus accumbens improved post-TBI auditory hallucinations, mood changes, and insomnia in a single female patient. Kuhn et al. reported a patient who had a substantial reduction in post- TBI self-mutilating behavior following posterior hypothalamus stimulation. An improvement in emotional adjustment and functional independence was reported in 4 TBI patients treated with nucleus accumbens DBS.Aside from the cognitive, psychiatric and mood improvements described above, DBS has also been investigated for the recovery of consciousness in patients in minimally conscious states. Out of 10 patients reported in the literature, an improvement was observed in 8 individuals using coma scales and related metrics.

Patients with memory and cognitive deficits following TBI that do not respond to conventional treatments experience a decrease in quality of life. Despite advances in neuroimaging, genetics, pharmacology and psychosocial interventions in the last half century, little progress has been made in altering the natural history of the condition or its outcome.

This study would explore whether a surgical therapy is safe and potentially effective in patients who develop refractory memory and cognitive deficits following TBI. Preclinical studies suggest that DBS may improve memory deficits in TBI models. Moreover, DBS delivered to the fornix has shown promising clinical results in patients with Alzheimer's disease. The main mechanism for the improvements induced by DBS in memory tests is the development of multiple forms of plasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male patients between age 18-70.
2. Diagnosis of memory and cognitive deficits in patients who suffered TBI will be defined according to the Diagnostic and Statistical Manual 5th edition (DSM-5).
3. Patients with cognitive disorder not otherwise specified, dementia, or amnestic disorder due to TBI will be considered.
4. Performance at least 1.5 standard deviations below the estimated premorbid intelligence (assessed by the American National Adult Reading Test) on memory tests (assessed by the California Verbal Learning Test; CVLT).
5. History of TBI for at least 1 year, preferably with evidence of failure to donepezil, cholinesterase inhibitors and cognitive therapy.
6. Ability to provide informed consent and comply with all testing, follow-ups and study appointments.

Exclusion Criteria:

1. Active neurologic disease, such as epilepsy or Alzheimer's disease.
2. Any contraindication to magnetic resonance imaging (MRI) scanning.
3. Presence of clinical and/or neurological conditions that may significantly increase the risk of the surgical procedure
4. Current suicidal or homicidal ideation.
5. Active neurologic disease, such as epilepsy.
6. Pregnancy.
7. Likely to relocate or move during the study's one year duration
8. Patients with renal dysfunction (GFR<60)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by SAFTEE | Every 2 weeks until the 8 weeks mark, every 4 weeks until 6 month mark and every two months until the 2 year mark
  The primary objective is to establish the safety of deep brain stimulation in a patient population with TBI and cognitive deficits using the Systematic Assessment for Treatment Emergent Events (SAFTEE)

CONTACTS AND LOCATIONS:
Overall Officials: Nir Lipsman, MD PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No